CLINICAL TRIAL: NCT05324813
Title: Examining Effects of Domain Specific Episodic Future Thinking on Cannabis Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Sofis (Industry)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Michael Sofis, Senior Scientist, Advocates for Human Potential
Organization: Advocates for Human Potential (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7420
Record Dates: First submitted 2022-03-16; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Marijuana Use; Marijuana Dependence; Tobacco Use; Alcohol Use, Unspecified
MeSH Terms: conditions — Marijuana Use; Marijuana Abuse; Tobacco Use; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Domain-Specific Episodic Future Thinking (Experimental)
  Interventions: Behavioral: Domain-Specific Episodic Future Thinking
- Episodic Recent Thinking Control Condition (Active Comparator)
  Interventions: Behavioral: Domain-Specific Episodic Future Thinking

INTERVENTIONS:
Behavioral: Domain-Specific Episodic Future Thinking — Individualized intervention that provides systematic prompts to enable creation and envisioning of positive future events across multiple life domains.

SUMMARY:
The overarching goal of this online study is to compare the efficacy of six (weekly) sessions of Domain-Specific Episodic Future Thinking (DS-EFT) relative an active control condition on improving the ability to value future rewards and reducing cannabis use (grams and days of use), tobacco use, and alcohol use among.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 or older
* reside in the U.S.
* report wanting to reduce cannabis use (4 or higher on scale of 1-10 with higher scores indicating greater desire to reduce use)
* report using cannabis at least 10 days in the last month
* report using cannabis at least 100 days in their lifetime
* Data quality checks passed

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of cannabis use grams | 1-week follow-up
Number of cannabis use days | 1-week follow-up

SECONDARY OUTCOMES:
Number of tobacco use days | 1-week follow-up
Number of alcohol use days | 1-week follow-up
Number of tobacco use times | 1-week follow-up
Number of alcoholic drinks | 1-week follow-up
Rate of delay discounting | 1-week follow-up
  5-trial adjusting delay discounting task

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Sofis, PhD, Principal Investigator — AHP
Locations (1):
- AHP Corporate Office, Sudbury, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol